CLINICAL TRIAL: NCT04872114
Title: A Prospective, Single-center, Open-label, Self Controlled Case Series Trial of Renal Sympathetic Denervation Using SyMapCath I™ Catheter and SYMPIONEER S1™ Stimulator/Generator for the Treatment of Hypertension in Patients on Hemodialysis (SMART-HD Trial)
Brief Title: Sympathetic Mapping/ Ablation of Renal Nerves Trial - Hemodialysis
Acronym: SMART-HD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: SyMap Medical (Suzhou), Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-12-HD
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Hypertension; Hemodialysis
MeSH Terms: conditions — Hypertension | interventions — Radionuclide Generators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal Sympathetic Denervation (Experimental): Percutaneous renal denervation using the SyMapCath I™ Catheter and SYMPIONEER S1™ Stimulator/Generator.
  Interventions: Device: SyMapCath I™ catheter and SYMPIONEER S1™ Stimulator/Generator

INTERVENTIONS:
Device: SyMapCath I™ catheter and SYMPIONEER S1™ Stimulator/Generator — Radiofrequency ablation of renal arterial sympathetic nerves

SUMMARY:
To evaluate the safety and efficacy of targeted renal sympathetic denervation using SyMapCath I™ in patients on hemodialysis with pharmacotherapy and uncontrolled hypertension for at least 6 months, then after standardized antihypertensive drug therapy (at least two drugs) for at least 28 days, office systolic blood pressure (BP) is still ≥ 150mmHg, ≤180mmHg.

DETAILED DESCRIPTION:
This is a prospective, single-center, open-label, self controlled case series trial, in which patients on maintenance hemodialysis are diagnosed with essential hypertension with at least six months of disease history and pharmacotherapy however their blood pressure still cannot be controlled. The patients will be informed, consent and get into a screening process. During the screening period patients will receive a standardized antihypertensive drug treatment for at least 28 days and office BP is still ≥ 150mmHg, ≤180mmHg, and meet the inclusion and exclusion criteria. These patients will conduct renal artery angiography followed by renal sympathetic nerve denvervation (30 patients). Patients with office BP which is not achieved ideal level (<140 mmHg) will titrate doses of classes of antihypertensive drugs according to a predefined standardized medication regimen until their office BP <140 mmHg.

Patients will be followed at 7 days after the procedure or at discharge from hospital, 1 month, 3 months and 6 months. Blood samples will be collected for drug tests to determine drug compliance of a patient.

Data collecting/management/statistical analysis and laboratory tests will be performed by independent, qualified organizations. Independent DSMB/CEC are formed and responsible for assessments of protocol deviations and natures of SAEs.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female subjects, 18≤age≤70;
2. Hemodialysis vintage ≥ 6 months, three sessions per week, and Kt/v≥1.0;
3. History of hypertension is longer than 6 months;
4. Average 24-hour ABPM systolic blood pressure ≥130 mmHg, or daytime systolic blood pressure ≥135 mmHg, or nocturnal systolic blood pressure ≥120 mmHg;
5. Office SBP ≥150mmHg and ≤180mmHg;
6. Patient with poor blood pressure control after 6 months of antihypertensive drug therapy, understands the purpose of this study, and is willing to participate and sign the Informed Consent; then the patient receives standard antihypertensive drug treatment (at least two drugs) for at least 28 days, drug compliance ≥80%, office BP ≥150 mmHg and ≤180 mmHg; Patient is compliant and willing to complete clinical follow-up.

Exclusion Criteria:

1. Renal artery anatomy is unqualified including: (1) diameter <4mm or treatable length <20mm; (2) Renal artery stenosis >50% or any renal artery aneurysms on either side; (3) History of renal artery PTA, including balloon angioplasty and stenting;
2. Average 24-hour systolic blood pressure (SBP) <135mmHg;
3. Pulse pressure > 80mmHg;
4. Using antihypertensive drugs, such as clonidine, minoxidil within 6 months;
5. Participated other clinical trials including both drug and medical device studies within 3 months enrollment;
6. Female with pregnant or lactating, or having plans for pregnancy within 1 year;
7. Patient with sleep apnea who needs chronic oxygen-breathing or mechanical ventilation support (for example, tracheostomy);
8. Patients previously or currently suffering from following diseases: (1) Essential pulmonary arterial hypertension; (2) Type I diabetes; (3) Severe cardiac valvular stenosis with contradictions to significantly reduce blood pressure; (4) History of myocardial infraction (MI), unstable angina, syncope or cerebrovascular accidents within half year; (5) History of primary aldosteronism, pheochromocytoma, aorta stenosis, hyperthyroidism or hyperparathyreosis; (6) Any disease conditions interfering the measurement of blood pressure (for instance, severe peripheral artery diseases, abdominal artery aneurysm, hemorrhagic disorders such as thrombocytopenia, hemophilia and severe anemia); (7) Plans to have surgery or cardiovascular interventions within following 6 months; (8) alcohol abuse or unknown drug dependence history; (9) Neuroticisms such as depression or anxiety disorders; (10) Non-compliant patients unable to finish the research per physician's requests;
9. Any contradictions to conduct renal artery stimulation and ablation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in office BP | 3 month after the treatment
  Reduction in office BP at 3 month after the treatment
The composite index of anti-hypertensive drugs | 6 months after the treatments
  The composite index of anti-hypertensive drugs at 6 months after the treatments

SECONDARY OUTCOMES:
Reduction in office BP | 1 month, 6 months
  Reduction in office BP at 1 month and 6 months after the treatment
Postoperative reduction in 24-hour Ambulatory Blood Pressure Monitoring (ABPM) reduction in systolic, diastolic and mean arterial blood pressure | 1 month, 3 months, 6 months
The control rates of reduction in office systolic blood pressure (SBP) by 10mmHg or Ambulatory Systolic Blood Pressure (ASBP) by 5mmHg | 1 month, 3 months, 6 months
The control rates of office systolic blood pressure ( SBP<140mmHg) | 6 month
  The control rates of office systolic blood pressure ( SBP<140mmHg) at 6 month after the treatment
Incidence of Intradialytic hypotension (IDH) | 1 month, 3 months, 6 months
  Decrease in systolic BP of ≥ 20 mm Hg during hemodialysis
All-cause death | 1 month, 3 months, 6 months
AEs, SAEs, and severe cardio-cerebrovascular events | 1 month, 3 months, 6 months
Success rate of the renal interventional therapy procedure | during the procedure
  the renal denervation catheter can be engaged to the correct position in renal artery, successfully performed renal nerve ablation procedure and has no related complications such as renal arterial perforation
Success rate of clinical treatment | 7 days after the procedure or at the time the patient is discharged from hospital
  based on succeed performance of renal interventional therapy procedure , there are no the procedure-related SAE, such as acute infection and renal dysfunction
Rate of renal artery stenosis assessed by CT angiography | 6 months
  stenosis > 70%

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided